CLINICAL TRIAL: NCT03239132
Title: MEditation for Post Stroke Depression
Acronym: MEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jennifer Beauchamp, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-SN-17-0583
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Depression
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breath-based meditation (Experimental): The experimental group will receive 4 group sessions of breath-based meditation over 4 weeks, as well as meditation educational materials.
  Interventions: Behavioral: Breath-based meditation; Behavioral: Meditation educational materials
- Control (Active Comparator): The control will receive meditation educational materials.
  Interventions: Behavioral: Meditation educational materials

INTERVENTIONS:
Behavioral: Breath-based meditation — The experimental group will receive 4 group sessions of breath-based meditation over 4 weeks.
  Arms: Breath-based meditation
Behavioral: Meditation educational materials — Meditation educational materials

SUMMARY:
The purpose of this study is to establish the feasibility and acceptability of a breath-based meditation in stroke survivors with post-stroke depression (PSD) and their informal caregivers, as well as to examine the effects of the breath-based meditation. The hypothesis is that the breath-based meditation will lead to decreases in the severity of symptoms of PSD, post-stroke anxiety (PSA), and post-traumatic stress disorder (PTSD), and decreases in plasma IL-1 pro-inflammatory cytokines post-intervention in stroke survivors with PSD and their informal caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors will be included if they speak English, can provide written informed consent, have a history of ischemic stroke, hemorrhagic, or transient ischemic attack within the past 8 weeks, have a Center for Epidemiologic Studies-Depression (CES-D) total score of 16 or greater suggestive of clinically significant depressive symptoms, and currently live at home.
* Informal caregivers will be included if they are speak English, can provide written informed consent, and self-identify as a first-time informal caregiver of a stroke survivor. -
* To reflect standard practice, stroke survivors and their informal caregivers will be eligible to participate in the study regardless of whether they are currently receiving anti-depressant medications; however, the dose must have been stable for at least one month prior to recruitment into the study.

Exclusion Criteria:

* Stroke survivors will be excluded if they currently reside outside of the home (e.g., rehabilitation center).
* Stroke survivors and their informal caregivers will be excluded if they have severe cognitive impairment (Montreal Cognitive Assessment (MoCA) cutoff score of 20), active psychosis, or bipolar disorder; if they currently abuse substances; or if they are acutely suicidal. Those currently receiving formal psychotherapy or currently engaging in self-identified meditation practices will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by number screened per week | 2 years
Feasibility as assessed by proportion of those eligible who enroll to the study | 2 years
Feasibility as assessed by number of participants who completed the study | 2 years
Feasibility as assessed by number of participants who adhered to the protocol | 2 years
Feasibility as assessed by number of participants who completed all study assessments | 2 years

SECONDARY OUTCOMES:
Post-Stroke Depression as assessed by the Center for Epidemiologic Studies Short Depression Scale (CES-D-R 10) | baseline, immediately after intervention ends, 4 weeks after intervention ends, 8 weeks after intervention ends
Post-Stroke Anxiety as assessed by the State-Trait Anxiety Inventory for Adults (STAI-AD) | baseline, immediately after intervention ends, 4 weeks after intervention ends, 8 weeks after intervention ends
Levels of plasma IL-1 family pro-inflammatory cytokines | baseline, immediately after intervention ends, 4 weeks after intervention ends, 8 weeks after intervention ends

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Sanner, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Beauchamp JES, Sharrief A, Chaoul A, Casameni Montiel T, Love MF, Cron S, Prossin A, Selvaraj S, Dishman D, Savitz SI. Feasibility of a meditation intervention for stroke survivors and informal caregivers: a randomized controlled trial. BMC Psychol. 2023 Jan 12;11(1):9. doi: 10.1186/s40359-022-01031-z. PMID 36635775